CLINICAL TRIAL: NCT03828864
Title: Pulsed Shortwave Therapy (PSWT) Chronic Low Back Pain
Brief Title: Pulsed Shortwave Therapy (ActiPatch®) Study in Chronic Low Back Pain
Acronym: PSWT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: BioElectronics Corporation (Industry)
Collaborators: Royal Prince Alfred Hospital, Sydney, Australia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: X18-0425
Record Dates: First submitted 2019-02-01; First posted 2019-02-04 (Actual); Last update posted 2019-02-05 (Actual); Status verified 2019-01

CONDITIONS: Chronic Low Back Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Active medical device and and identical dummy device (placebo) that does not emit the pulsed shortwave signal.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Active Pulsed Shortwave therapy (Active Comparator): Application of the medical device emitting pulsed shortwave therapy. The medical device is used over the site of pain.
  Interventions: Device: Pulsed Shortwave Therapy
- Placebo Pulsed Shortwave therapy (Placebo Comparator): Application of the medical device that does not emit pulsed shortwave therapy. The medical device is used over the site of pain.
  Interventions: Device: Placebo Pulsed Shortwave Therapy

INTERVENTIONS:
Device: Pulsed Shortwave Therapy — Pulsed Shortwave Therapy device placed over the site of pain for 16 hrs per day
  Other Names: ActiPatch
  Arms: Active Pulsed Shortwave therapy
Device: Placebo Pulsed Shortwave Therapy — Placebo Pulsed Shortwave Therapy device placed over the site of pain for 16 hrs per day
  Other Names: Placebo ActiPatch
  Arms: Placebo Pulsed Shortwave therapy

SUMMARY:
This study aims to test the efficacy of the ActiPatch® device by means of a randomized double blind controlled trial in a convenience sample of chronic low back pain patients at RPAH pain clinic. Outcome measures are validated psychometric measures evaluating known determinants of pain related disability, functional capacity measures, and pain scores; and a bespoke questionnaire assessing fidelity with recommended usage, and willingness to reduce analgesic or other pain related medications with the future assistance of the ActiPatch®.

DETAILED DESCRIPTION:
This study aims to test the efficacy of the ActiPatch® device by means of a randomised double blind controlled trial in a convenience sample of chronic low back pain patients at Royal Prince Alfred Hospital (RPAH) pain clinic. Outcome measures are validated psychometric measures evaluating known determinants of pain related disability, functional capacity measures, and pain scores; and a bespoke questionnaire assessing fidelity with recommended usage, and willingness to reduce analgesic or other pain related medications with the future assistance of the ActiPatch®.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the trial.
* In the Investigator's opinion, is able and willing to comply with all trial requirements.
* Male or female ages 18 or above with stable chronic lower back pain
* Females of childbearing must be on birth control or practice abstinence during the study period.
* In the event of possible pre-existing pregnancy, women of childbearing age will be screened with a urine pregnancy test. Women of childbearing potential are defined as any female who has experienced menarche and who is not permanently sterile or postmenopausal. Postmenopausal is defined as 12 consecutive months with no menses without an alternative medical cause.
* ≥3 months duration of chronic low back pain i.e. cut off period for acute pain
* a current BPI pain rating ≥5/10 on one of the 4 of the four pain VAS scales on the BPI
* Most of the pain in the body is present in the lower back or buttock, NOT in the lower extremities, as determined during screening by the principal investigator. The investigator will verbally ask the participant if most of the pain being experienced is in the lower back/buttock area, and rely on the response for inclusion into the study.
* Able to complete and tolerate treatment for the study period.
* Pain stable in one area of the low back- i.e. not variable in location
* Medication regime stable over the last 3 months

Exclusion Criteria:

* Female participant who is pregnant.
* Subjects using personal home based electrical stimulation devices
* Prior home use of pulsed shortwave therapy. i.e ActiPatch®
* Scheduled elective surgery or other procedures requiring general anaesthesia during the trial.
* Planned or scheduled variation in pain related medication (analgesic or psychoactive) regime during the course of the trial.
* Active psychiatric disorders (e.g. participants using antipsychotic medication, with bipolar disorder or schizophrenia).
* Subjects with other concomitant illnesses (e.g., malignancy) which, in the opinion of the investigator, would preclude successful subject participation
* Subjects diagnosed with a history of significant mood disorder will be excluded (Note that subjects with depression or anxiety with adequate control would be acceptable). Participants would be required to be stable with their moods (EPPOC data or psychological or psychiatric evaluation can be referenced in the case of doubt)
* Any other significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the trial, or may influence the result of the trial, or the participant's ability to participate in the trial.
* Participants who have participated in another research trial involving an investigational product in the past 12 weeks
* Participants who are planning to change any other variables during the study period likely to affect their pain or function e.g. commencement of an exercise class; ceasing allied health treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Estimated)
Dates: Start 2019-02-01 (Estimated); Primary Completion 2020-02-01 (Estimated); Study Completion 2020-05-01 (Estimated)

PRIMARY OUTCOMES:
Brief Pain Inventory (BPI) Short Form | 30 days
  The BPI-SF is a questionnaire - self-administered or by interview - that assesses both pain intensity and pain interference in common aspects of one's life. It has reliability & validity across cultural and language groups & is one of the standard measures used by the national Electronic Persistent Pain Outcomes Collaboration (ePPOC) that collates data from various Pain Management Centres to evaluate outcomes in pain clinics Australia wide.
  Scoring
  Question answers are complied into two categories:
  1. Pain severity is 0 - 10, with 10 being worst pain possible
  2. Pain inference score is 0 - 10, with 10 being worst possible pain inference

SECONDARY OUTCOMES:
Central Sensitisation Inventory - short form (CSI-9) | 30 days
  Central Sensitisation (CS) is thought to be one underlying mechanism for the prevalence of chronic pain and the ActiPatch® device is believed to reduce central sensitization. Use of the CSI-9 will be used to assess the extent to which central sensitization is present in the study cohort and if use of the device produces a change in CS. This will then allow appraisal of the role of central sensitization in any outcomes achieved.
  Scoring, scores are totaled from the assessment Five severity levels (subclinical = 0-29, mild = 30-39, moderate = 40-49, severe = 50-59, and severe = 60-100) central sensitization
Pain Sleep Questionnaire (PSQ-3) Scoring 0-30 0 no sleep disturbance and 30 worst sleep disturbance | 30 days
  The interaction between sleep disturbance and chronic pain is widely reported in the literature, and is thought to be a two way interaction. Use of the PSQ-3 will be used to assess the extent to which perceived sleep disturbance is present in the study cohort and if use of the ActiPatch® device is associated with a change in sleep quality. Addressing sleep quality may help to treat chronic pain including LBP and thereby have clinical treatment applications.
  Scoring 0-30, 0 no sleep disturbance and 30 worst sleep disturbance Three visual analog scales of 0-10

CONTACTS AND LOCATIONS:
Overall Officials: Graeme Campbell, Principal Investigator — Royal Prince Alfred Hospital, Sydney, Australia; Arun Aggarwal, Professor, Study Chair — Royal Prince Alfred Hospital, Sydney, Australia

IPD SHARING:
Plan to Share IPD: No